CLINICAL TRIAL: NCT05462574
Title: Clinical and Mechanistic Understanding of Right Ventricular Steatosis in Pulmonary Arterial Hypertension (PAH)
Brief Title: Right Ventricle Lipid in Pulmonary Arterial Hypertension (PAH)
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Evan Brittain, Associate Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: 221138; HL155278 (Other Grant/Funding Number: NHLBI)
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension; Heritable Pulmonary Arterial Hypertension; Pulmonary Arterial Hypertension Associated With Connective Tissue Disease
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Pulmonary Arterial Hypertension (PAH): Participants with heritable, idiopathic, and scleroderma associated PAH.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The investigators propose to study the relationship between right ventricle (RV) steatosis and RV function, exercise capacity, and outcomes in humans with pulmonary arterial hypertension (PAH) and to identify potential drivers of lipid accumulation.

DETAILED DESCRIPTION:
The investigators propose to test the hypothesis that abnormal lipid metabolism in PAH leads to delivery of fatty acids in excess of RV oxidative capacity, resulting in steatosis and lipotoxicity. The objectives of the study are to: 1) Define the relationships between RV steatosis, RV function, and exercise capacity; 2) Identify mechanistic drivers of RV steatosis including BMPR2 expression and lipid metabolism; 3) Examine lipid metabolism in PAH skeletal muscle as a potential driver of reduced functional capacity.

In Aim 1 (clinical relevance) the investigators will measure RV and left ventricle (LV) lipid in participants with heritable, idiopathic, and scleroderma- associated PAH. Participants will undergo the 6-minute walk test, cardiopulmonary exercise testing, and will be followed for clinical events. A subgroup will undergo repeat MRS at four timepoints over three years to determine the natural history of steatosis.

In Aim 2 (mechanism), the investigators will perform metabolomic/lipidomic profiling of peripheral and coronary sinus plasma and measure BMPR2 expression to identify potential drivers of steatosis.

In Aim 3 (specificity), the investigators will perform MRS on skeletal muscle in Aim 1 participants and matched healthy controls to clarify the systemic effects of lipid metabolic defects in PAH.

ELIGIBILITY:
Inclusion criteria:

* ≥ 18 years old
* Diagnosed with idiopathic, heritable, connective tissue disease-associated PAH, associated pulmonary arterial hypertension (PAH), or drug-or toxin-associated PAH according to World Health Organization (WHO) consensus recommendations.
* Stable PAH-specific medication regimen for three months prior to enrollment. Adjustments in IV prostacyclin for side effect management are allowed. Diuretic adjustments are permitted.
* WHO Functional Class I-III
* Ambulatory
* Able to have an MRI/MRS, perform a 6MWD test, and cardiopulmonary exercise test

Exclusion criteria:

* Pregnancy
* Diagnosis of PAH etiology other than idiopathic, heritable, connective tissue disease - associated PAH or associated with drugs and toxins
* WHO Functional class IV heart failure
* Requirement for continuous oxygen
* Unable to have an MRI/MRS, perform a 6MWD test, or cardiopulmonary exercise test.
* Patients with implanted/embedded ferromagnetic material that would preclude cardiac MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PAH will be recruited from the Center for Pulmonary Vascular Disease (CPVD) at Vanderbilt University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Right Ventricular (RV) Ejection Fraction | Baseline to 36 months
  Change in RV ejection fraction will be measured by cardiac MRI.
Change in Right Ventricular (RV) Lipid Content | Baseline to 36 months
  Change in RV lipid content will be measured by cardiac proton magnetic resonance spectroscopy (MRS). Lipid content is expressed as a percent of the voxel occupied by lipid.
Identification of metabolic markers (dihyroxybutyrate, acetylputriscene, hydroxystearate and glucuronate) in the peripheral circulation and coronary sinus. | Baseline to 36 months
  Metabolite markers will be measured by ultrahigh performance liquid chromatography and mass spectrometry.
Ratio of BMPR2 isoform B/A. | Baseline to 36 months
  BMPR2 isoforms A and B and wild type gene expression will be measured by real-time polymerase chain reaction (PCR) and validated by measuring protein content using Western blot test.
Change in skeletal muscle lipid content. | Baseline to 36 months
  Change in skeletal muscle lipid content will be measured by skeletal muscle proton MRS. Lipid content is expressed as percent triglyceride (%TG)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Brittain, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States